CLINICAL TRIAL: NCT02766972
Title: Rapid Ventricular Pacing in Surgical Treatment of Intracranial Aneurysms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Clinic Frankfurt (Other)
Responsible Party: Principal Investigator, Juergen Konczalla, MD, University Clinic Frankfurt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 497/13
Record Dates: First submitted 2016-04-29; First posted 2016-05-10 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Intracranial Aneurysm; Surgical Clip
Keywords: Intracranial Aneurysm; Surgical Clipping; Rapid Ventricular Pacing
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RVP (Experimental)
  Interventions: Procedure: Rapid Ventricular Pacing

INTERVENTIONS:
Procedure: Rapid Ventricular Pacing — Use of Rapid Ventricular Pacing to improve surgical clipping of intracranial aneurysms

SUMMARY:
Treatment of complex unruptured intracranial aneurysms (UIA) remains challenging to date. Therefore, advanced techniques are required to achieve an optimal result in treating these patients safely. In this study, the safety and efficacy of rapid ventricular pacing (RVP) to facilitate microsurgical clip-reconstruction has been studied prospectively in a joined neurosurgical, anesthesiological and cardiological study.

DETAILED DESCRIPTION:
Treatment of complex unruptured intracranial aneurysms (UIA) remains challenging to date. Therefore, advanced techniques are required to achieve an optimal result in treating these patients safely. In this study, the safety and efficacy of rapid ventricular pacing (RVP) to facilitate microsurgical clip-reconstruction has been studied prospectively in a joined neurosurgical, anesthesiological and cardiological study. Patients with complex UIA were prospectively enrolled and the safety and efficacy of RVP were evaluated recording cardiovascular events and outcome of the patients as well as the amount of aneurysm occlusion after the surgical clip-reconstruction procedure.

ELIGIBILITY:
Inclusion Criteria:

* complex UIA intended to be treated by microsurgical clip-reconstruction
* application of RVP intra-operatively

Exclusion Criteria:

* structural heart disease or conductance abnormalities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
modified Rankin scale | 6 months

SECONDARY OUTCOMES:
Efficacy of flow reduction and improvement of clip application | intraoperatively
  Efficacy of flow reduction (failure rate of pacing; measuring of heart rate and blood pressure).
  Also improvement of clip application: performing surgeon has to complete a questionnaire.
safety of pacing catheter | intraoperatively upt o 24 hours after operation
  Complications during insertion, positioning, application (intraoperatively) and removal of pacing catheter (postoperatively on ICU). Anesthesiologist has to complete a questionnaire.
Cardiovascular events | intraoperatively upt o 24 hours after operation
  All cardiovascular events will be documented (like arrhythmias etc.). Also preoperative heart values (of Troponin T, CK, CK-MB) and values after operation and one day after operation will be documented and afterwards analyzed.
  Reference values (05/2016): CK <190 U/l; CK-MB <24 U/l; Troponin T <14pg/ml Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment were documented and analyzed.
occlusion rate of aneurysm | 1 week after operation
  Angiography to control the occlusion of the aneurysm, regularly 1 week after surgical clipping.

CONTACTS AND LOCATIONS:
Locations (1):
- Goethe University Hospital, Frankfurt am Main, Germany

REFERENCES:
- [Derived] Konczalla J, Platz J, Fichtlscherer S, Mutlak H, Strouhal U, Seifert V. Rapid ventricular pacing for clip reconstruction of complex unruptured intracranial aneurysms: results of an interdisciplinary prospective trial. J Neurosurg. 2018 Jun;128(6):1741-1752. doi: 10.3171/2016.11.JNS161420. Epub 2017 Aug 18. PMID 28820303